CLINICAL TRIAL: NCT00144547
Title: An Open-label, Extension, Phase III Study to Evaluate the Long-term Safety and Efficacy of MRA in Patients With RA Who Participated in Study MRA012JP
Brief Title: Long-term Treatment Study of MRA for Rheumatoid Arthritis (RA) From Study MRA012JP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRA214JP
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MRA(Tocilizumab)

INTERVENTIONS:
Drug: MRA(Tocilizumab) — 8mg/kg(i.v.)/4weeks

SUMMARY:
This is an open-label, extension, Phase III study to evaluate the long-term safety and efficacy of MRA in patients with RA who participated in Study MRA012JP.

ELIGIBILITY:
Inclusion criteria

* Patients must suffer from RA, and must have participated in the preceding study.
* Patients must have been confirmed to be appropriate on week 52 of the preceding study by X radiography.

Exclusion criteria

* Patients evaluated as belonging to Steinbrocker's class IV within 4 weeks before administration of the study drug
* Patients who have not been registered by 3 months after week 52 of the preceding study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2004-04; Primary Completion 2008-08 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Patients fron MRA Group of previous study:The frequency of amelioration of at least 20% in terms of the ACR criteria compared to the beginning of the treatment in previous study(MRA012JP) | 0W,4W,8W,12W,LOBS
Patients fron non-MRA Group of previous study:The frequency of amelioration of at least 20% in terms of the ACR criteria | 0W,4W,8W,12W,LOBS

SECONDARY OUTCOMES:
Time courses of DAS28, frequencies of amelioration of at least 20%, 50%, and 70% in terms of the ACR criteria, each item in the ACR core set | 0W,4W,8W,12W,LOBS
Frequency, severity, and seriousness of adverse events and adverse drug reactions | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Takahiro Kakehi, Study Director — Chugai Pharmaceutical